CLINICAL TRIAL: NCT00353821
Title: Cytokine Gene Polymorphisms in Allotransplant Donors
Brief Title: Investigating Cytokine Genes of Stem Cell Donors
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030201; 03-H-0201
Record Dates: First submitted 2006-07-18; First posted 2006-07-19 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2018-03-02

CONDITIONS: Stem Cell Transplantation
Keywords: Tumor Necrosis Factor Alpha (TNF-Alpha); Interferon-Gamma (IFN-Gamma); Interleukin-10 (IL-10); Interleukin-6 (IL-6); Interleukin-1 (IL-1 Ra); Interleukin-1 Receptor Antagonist (IL-1 Ra); Vitamin D Receptor (VitD R)

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study seeks to investigate the factors that may account for the differences in the way a stem cell recipient s immune system works after a transplant. It will focus on cytokine genes, which give specific instructions to the genes and which may influence immune system response. More specifically, the purpose of the study is to find out how gene polymorphisms (gene variations among the population) affect the success or failure of a stem cell transplant.

Study participants will have donated blood for a stem cell transplant. They will be asked to give consent for NIH personnel to run special tests on these blood samples, which will have been placed in storage. It is hoped that blood samples will be studied from 600 stem cell donors.

DETAILED DESCRIPTION:
The NHLBI Stem Cell Allotransplantation Program is researching methods to improve allogeneic stem cell transplantation. We are particularly interested in identifying factors, which result in individual variability in outcomes. Cytokines are biological modulators of the immune system known to influence various phases of the immune response. Normal variations in the genetic material coding for cytokines (Cytokine Gene Polymorphisms or CGPs) are believed to account for some of the differences in the inflammatory response between individuals. In the future, we hope to tailor stem cell transplantation to take into account these immunological profiles. In order to characterize the effect of any such intervention, we first need to better understand the role CGPs play in immune responses in normal, healthy persons. This involves testing for the presence or absence of a polymorphism in healthy individuals, and comparing with a validated in vitro assay. None of these polymorphisms are associated with known clinical disease to be classifiable as a 'genetic defect'. Moreover, we will not correlate these polymorphisms with clinical studies to identify traits in the sample donors. We plan to utilize stored blood samples from stem cell transplant donors who have previously participated on a hematology branch protocol as well as consent future donors.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participation as a stem cell donor on a Hematology Branch protocol.

For adults: Ability to comprehend the investigational nature of the study and provide informed consent. For minors: Written informed consent from one parent or guardian. Informed assent from minors: The process will be explained to the minor on a level of complexity appropriate for their age and ability to comprehend.

Age greater than or equal to 2 and less than or equal to 80.

EXCLUSION CRITERIA:

Subjects unable to comprehend the investigational nature of the laboratory research.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-06-05; Study Completion 2018-03-02

CONTACTS AND LOCATIONS:
Overall Officials: A. John Barrett, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Socie G, Loiseau P, Tamouza R, Janin A, Busson M, Gluckman E, Charron D. Both genetic and clinical factors predict the development of graft-versus-host disease after allogeneic hematopoietic stem cell transplantation. Transplantation. 2001 Aug 27;72(4):699-706. doi: 10.1097/00007890-200108270-00024. PMID 11544434
- [Background] Cavet J, Middleton PG, Segall M, Noreen H, Davies SM, Dickinson AM. Recipient tumor necrosis factor-alpha and interleukin-10 gene polymorphisms associate with early mortality and acute graft-versus-host disease severity in HLA-matched sibling bone marrow transplants. Blood. 1999 Dec 1;94(11):3941-6. PMID 10572111
- [Background] Cavet J, Dickinson AM, Norden J, Taylor PR, Jackson GH, Middleton PG. Interferon-gamma and interleukin-6 gene polymorphisms associate with graft-versus-host disease in HLA-matched sibling bone marrow transplantation. Blood. 2001 Sep 1;98(5):1594-600. doi: 10.1182/blood.v98.5.1594. PMID 11520812